CLINICAL TRIAL: NCT06048679
Title: Is Reducing Flow in Affected Branch Pulmonary Arteries in Patients With Partial Anomalous Pulmonary Venous Drainage Using a Percutaneous Approach Safe and Efficacious? - a Pilot Study
Brief Title: Percutaneous Treatment of Partial Anomalous Pulmonary Venous Drainage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PA22/149367
Record Dates: First submitted 2023-08-24; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Partial Anomalous Pulmonary Venous Connection
Keywords: congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- main (Other)
  Interventions: Device: Endovascular pulmonary artery flow-limiting covered stent implantation

INTERVENTIONS:
Device: Endovascular pulmonary artery flow-limiting covered stent implantation — selective reduction of flow in the pulmonary arteries affected by anomalous pulmonary venous drainage using a modified flow-limiting covered stent

SUMMARY:
Partial anomalous pulmonary venous drainage (PAPVD) occurs in around 1 in every 1000 people. Blood from part of the lung returns to the wrong side of the heart, causing the heart to stretch. This causes breathlessness and heart rhythm problems in later life. PAPVD can currently only be fixed by open heart surgery, and when the abnormality affects the right lung, even this can be impossible.

This study is designed to examine whether a new keyhole procedure to limit blood flow through the affected lung segments can be safely used to reduce the impact of PAPVD on the heart, reducing symptoms, protecting against heart rhythm problems, and avoiding the need for open heart surgery.

In this study, a flow limiting device will be positioned in the affected lung artery to reduce blood flow to this segment of lung. The procedure is performed under a general anaesthetic, and is done either as a day case or a single overnight stay in hospital. X-rays are used to guide the positioning of the stent. The procedure is performed as a keyhole procedure through a 3 mm cut in the groin.

The investigators will use heart ultrasound, heart MRI and exercise testing before and six months after the procedure to assess the safety and effect of the flow limiter.

The flow limitation device will either be a standard covered stent used in every day practice, but with a modified balloon for deployment, a vascular plug or similar vascular occlusion device which can be modified to restrict rather than occlude flow. If there is a problem with the flow limitation being too severe, the stent can be fully inflated returning the flow back to normal, and the vascular plug can be retrieved using another key hole procedure.

DETAILED DESCRIPTION:
PAPVD has been reported in 0.2% of the population undergoing CT scans and in 0.4 - 0.7% of the population in autopsy studies. They can be associated with superior sinus venosus atrial septal defects or can be present in isolation.

PAPVD causes blood which should be draining from the lungs into the left hand side of the heart to drain into the right side of the heart. Thus PAPVD results in a left to right shunt of varying proportions dependent upon the number of lobes involved. Long term sequelae reflect the impact of the resultant volume loading of the right heart, which can lead to atrial arrhythmia and right heart failure in later life and these patients can develop pulmonary hypertension. Patients with significant left to right shunts often present with symptoms of breathlessness and poor exercise tolerance, which worsen as they age.

Historically, PAPVD has only been considered suitable for surgical repair. This requires an open heart procedure, including cardio-pulmonary bypass, and necessitates around a week in hospital, and a three month recovery period. Surgical repair is technically challenging due to anatomical considerations, particularly in right sided anomalous veins, and there is a relatively high risk of pulmonary venous thrombosis post operatively due to low velocity venous flow. Current European Society of Cardiology guidelines recommend that technical suitability for repair and operative risk must be weighed against the potential benefit of intervention. These guidelines also state that it is unusual for a single anomalous pulmonary venous connection of only one pulmonary lobe to result in a sufficient volume load to justify the risk of surgical repair.

ELIGIBILITY:
Inclusion Criteria:

* Haemodynamically & Functionally significant PAPVD (all of the following)

  * Right heart dilated on trans thoracic echo
  * cardiac MRI Qp:Qs ≥ 1.3:1, and right ventricular to left ventricular volume (RV:LV) ratio ≥ 1.5:1
  * Maximal oxygen consumption (VO2 max) on cardiopulmonary exercise testing < 85% predicted
  * Normal pulmonary artery pressure
* No contra-indication to pulmonary artery intervention procedure under general anaesthetic
* Able to give informed consent

Exclusion Criteria:

* Contra-indication to cardiac MRI
* Not able to give informed consent
* Contra-indication to pulmonary artery intervention under general anaesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Right ventricular end diastolic volume | 6 months post procedure
  changes in right ventricular end diastolic volume assessed by MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haramati LB, Moche IE, Rivera VT, Patel PV, Heyneman L, McAdams HP, Issenberg HJ, White CS. Computed tomography of partial anomalous pulmonary venous connection in adults. J Comput Assist Tomogr. 2003 Sep-Oct;27(5):743-9. doi: 10.1097/00004728-200309000-00011. PMID 14501365
- [Background] HEALEY JE Jr. An anatomic survey of anomalous pulmonary veins: their clinical significance. J Thorac Surg. 1952 May;23(5):433-44. No abstract available. PMID 14928263
- [Background] Hegde M, Manjunath SC, Usha MK. Isolated Partial Anomalous Pulmonary Venous Connection: Development of Volume Overload and Elevated Estimated Pulmonary Pressure in Adults. J Clin Imaging Sci. 2019 Jun 14;9:29. doi: 10.25259/JCIS-8-2019. eCollection 2019. PMID 31508264
- [Background] Lewis RA, Billings CG, Bolger A, Bowater S, Charalampopoulos A, Clift P, Elliot CA, English K, Hamilton N, Hill C, Hurdman J, Jenkins PJ, Johns C, MacDonald S, Oliver J, Papaioannou V, Rajaram S, Sabroe I, Swift AJ, Thompson AAR, Kiely DG, Condliffe R. Partial anomalous pulmonary venous drainage in patients presenting with suspected pulmonary hypertension: A series of 90 patients from the ASPIRE registry. Respirology. 2020 Oct;25(10):1066-1072. doi: 10.1111/resp.13815. Epub 2020 Apr 6. PMID 32249494
- [Background] Geva T, Martins JD, Wald RM. Atrial septal defects. Lancet. 2014 May 31;383(9932):1921-32. doi: 10.1016/S0140-6736(13)62145-5. Epub 2014 Apr 8. PMID 24725467
- [Background] Stewart RD, Bailliard F, Kelle AM, Backer CL, Young L, Mavroudis C. Evolving surgical strategy for sinus venosus atrial septal defect: effect on sinus node function and late venous obstruction. Ann Thorac Surg. 2007 Nov;84(5):1651-5; discussion 1655. doi: 10.1016/j.athoracsur.2007.04.130. PMID 17954078
- [Background] Baumgartner H, De Backer J, Babu-Narayan SV, Budts W, Chessa M, Diller GP, Lung B, Kluin J, Lang IM, Meijboom F, Moons P, Mulder BJM, Oechslin E, Roos-Hesselink JW, Schwerzmann M, Sondergaard L, Zeppenfeld K; ESC Scientific Document Group. 2020 ESC Guidelines for the management of adult congenital heart disease. Eur Heart J. 2021 Feb 11;42(6):563-645. doi: 10.1093/eurheartj/ehaa554. No abstract available. PMID 32860028